CLINICAL TRIAL: NCT02958254
Title: Ultrasound Measurements of Hamstring Muscles Thickness Are a Valid Tool
Brief Title: Ultrasound Measurements Hamstring Muscles Thickness
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Josep C. Benitez Martinez, Associate Professor, University of Valencia
Other Study IDs: H1458067703008
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Muscle Injury; Muscle Atrophy
Keywords: hamstring; ultrasonography; validation; magnetic resonance imaging; muscle thickness
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
No previous studies have compared the association between muscle thickness (MT) and muscle cross-sectional area (CSA) in healthy volunteers. The main aim of this study is to investigate the validity of ultrasound in assessing the muscle thickness of hamstrings muscle.

Study design:

A cross-sectional-validity study.

Setting:

University

Participants:

X football players of an amateur football team (X healthy volunteers and X patients with a previous hamstring injury).

DETAILED DESCRIPTION:
X healthy volunteers, from an amateur football team, and X football players with previous history of hamstring injury from an orthopaedic clinic, comprised the subjects in this study. Hamstring muscle injury was defined as "a traumatic distraction or overuse injury to the hamstring muscle leading to a player being unable to fully participate in training or match play".

The Control Group (CG) were healthy, had neither surgery/trauma in their lower extremities, nor history of hamstring injury, and there were no abnormal findings in their physical examination. The exclusion criteria included participants who: (1) had metal implants or pace makers, (2) weighted more than 200 kg (MRI table limitations), and (3) were unable to complete testing. In the Injured Group, patients were also excluded if their previous injury was originated from a non-muscular source (e.g., inguinal or femoral hernia, nerve entrapment, lumbosacral pathology), or if still had symptoms, had not returned to practice and had not been participating in track and field since their last injury.

The Study Group (SG) had history and diagnosis of hamstring injury assessment with diagnosis image technique (ultrasound or MRI), and at least 2 of the next criteria: 1. When the injury happened disability to practise with the team at least one week; 2. Lost at least one match; 3. Felt pain when trying to kick the ball or run fast; 4. Receive specific treatment (medical or physiotherapy) for the injury; 5. Needed a period plan to return to play.

Participants were screened for contraindications to MRI before ultrasound assessment and an MRI scan of the hamstring muscles of both legs were performed. MRI was performed within 24 h of the ultrasound scan. The subjects were instructed not to consume alcohol or perform any moderate to heavy exercise for 24 hours prior to each imaging session.

Muscle thickness was defined as the distance between the bone-muscle interface and the adipose tissue-muscle interface. The measurement was made from the most superficial edge of the bright line representing the interface of the bony cortex and the muscle to the most superficial edge of the bright line representing the interface of the outer fascial layer of the muscle and the subcutaneous adipose tissue. When the bone was not in contact of the muscle the two fascial layer were used.

ELIGIBILITY:
Inclusion Criteria:

* Practice at least twice per week
* Playing soccer more than 5 years
* Inform Consent signed

Exclusion Criteria:

* 18 years or older
* Had metal implants or pace makers
* Weighted more than 200 kg (MRI table limitations)
* Were unable to complete testing

Injuries players:

* History and diagnosis of hamstring injury
* Assessment with diagnosis image technique (ultrasound or MRI)
* At least 2 of the next criteria:

  1. When the injury happened disability to practise with the team at least one week;
  2. Lost at least one match
  3. Felt pain when trying to kick the ball or run fast
  4. Receive specific treatment (medical or physiotherapy) for the injury
  5. Needed a period plan to return to play

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers from an amateur soccer team
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2021-04-26 (Actual); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Hamstring muscles thickness in millimeters by Ultrasound | 30 minutes
Hamstring muscles thickness in millimeters by Magnetic Resonance Image | 1 hour

SECONDARY OUTCOMES:
Cross-Sectional Area of the hamstring muscles in square millimeters by Ultrasound | 30 minutes
Cross-Sectional Area of the hamstring muscles in square millimeters by Magnetic Resonance Image | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Josep Benítez-Martínez, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ekstrand J, Hagglund M, Walden M. Epidemiology of muscle injuries in professional football (soccer). Am J Sports Med. 2011 Jun;39(6):1226-32. doi: 10.1177/0363546510395879. Epub 2011 Feb 18. PMID 21335353